CLINICAL TRIAL: NCT02875184
Title: Observational Study of Apremilast Use and Effectiveness in Patients With Psoriatic Arthritis in The Netherlands
Brief Title: A Study of Apremilast Use and Effectiveness in Patients With Psoriatic Arthritis in The Netherlands
Acronym: REWARD
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-10004-PSA-009; CC-10004-PSA-009-20200071 (Other: Amgen)
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Arthritis, Psoriatic
Keywords: Psoriatic Arthritis; Apremilast; CC-10004
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Psoriatic arthritis patients treated with apremilast: Psoriatic arthritis patients who are treated with apremilast according to daily practice

SUMMARY:
This is a multicenter, prospective, non-interventional, observational single arm study.

100 patients will be recruited in the Netherlands over a one year period. In all cases, the decision to treat the patient with apremilast will be made prior to the decision to enter the subject into this study. Treatment will be according to routine clinical practice and based on recommendations as per the Summary of Product Characteristics (SPC) of apremilast (Otezla®). Each patient will be followed up for a maximum of 24 months.

DETAILED DESCRIPTION:
The objective of this non-interventional study is to describe patient reported outcomes, effectiveness and real-life use of apremilast treatment in patients with psoriatic arthritis (PsA).

ELIGIBILITY:
Inclusion Criter

* Patients ≥ 18 years of age who understand and voluntarily sign an informed consent form.
* Patients starting treatment with apremilast for psoriatic arthritis.

Exclusion Criteria:

* Refusal to participate in the study.
* Language barrier for completing the questionnaires.
* Women who are pregnant or breast-feeding.
* Hypersensitivity to the active substance or to any of the excipients.
* Prior exposure to apremilast
* Initiation of apremilast treatment by a dermatologist for psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two hundred adult patients treated with apremilast for psoriatic arthritis will be recruited. In all cases, the decision to treat the patient with apremilast will be made prior to the decision to enter the subject into the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a Health Assessment Questionnaire - Disability Index (HAQ-DI) score of ≤ 0.5 or with a decrease of ≥ 0.3 of the HAQ-DI score compared with baseline | Up to 24 months
  The HAQ is a general questionnaire to assess physical functioning.

SECONDARY OUTCOMES:
Change from Baseline in Psoriatic Arthritis Impact of Disease (PsAID) at various time point | Up to 24 months
  PsAID is a general questionnaire that measures the health impact of psoriatic arthritis.
Change from Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM) at various time points | Up to 24 months
  The TSQM questionnaire is a general measure of treatment satisfaction across medication types and patient conditions.
Change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at month 6 | Up to 6 months
  The BASDAI is used for measuring and evaluating disease activity in Ankylosing Spondylitis.
Change from Baseline in Dermatology Life Quality Index (DLQI) at month 6 | Up to 6 months
  The DLQI is a dermatology specific Quality of Life instrument.
Change from Baseline in Short Form 36 (SF36) at 12 months | Up to 12 months
  The SF-36v2® Health Survey measures functional health and well-being from the patients point of view. It can be used across age (18 and older), disease and treatments.
Change from Baseline in EuroQol-5 dimensions (EQ5D) at 12 months | Up to 12 months
  EQ-5D is a standard instrument to measure of health status.
Change from Baseline in visual analogue scales (VAS) at various time point | Up to 24 months
  VAS is a simple assessment of the global health, itch and pain severity using a visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (20):
- Netherlands (20):
  - Reumazorg ZWN, Lelystad/Emmeloord, Flevoland
  - St. Jansdal, Harderwijk, Gelderland
  - Viecuri Medisch Centrum, Venlo, Limburg
  - Amphia, Breda, North Brabant
  - Elkerliek ziekenhuis, Helmond, North Brabant
  - Reumazorg ZWN, Roosendaal, North Brabant
  - MC Leeuwarden, Leeuwarden, Provincie Friesland
  - Beatrix Ziekenhuis, Gorinchem, South Holland
  - Groene Hart Ziekenhuis, Gouda, South Holland
  - Erasmus MC, Rotterdam, South Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - Reumazorg ZWN, Goes, Zeeland
  - Research Site, Breda
  - Research Site, Gorinchem
  - Research Site, Gouda
  - Research Site, Harderwijk
  - Research Site, Leeuwarden
  - Research Site, Roosendaal
  - Research Site, Rotterdam
  - Research Site, Venlo

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Expanded Access for CC-100004 — https://clinicaltrials.gov/ct2/show/NCT02875184?term=CC-10004-PSA-009&rank=1